CLINICAL TRIAL: NCT00000389
Title: Research Unit on Pediatric Psychopharmacology Anxiety Treatment Study
Brief Title: Treatment for Anxiety in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Masking: Double | Purpose: Treatment
Other Study IDs: N01 MH60005; N01 MH60016; DSIR CT
Record Dates: First submitted 1999-11-02; First posted 1999-11-03 (Estimated); Last update posted 2007-06-14 (Estimated); Status verified 2005-11

CONDITIONS: Obsessive-Compulsive Disorder; Anxiety Disorders; Generalized Anxiety Disorder; Social Phobia; Separation Anxiety
Keywords: Adolescence; Anxiety Disorders; Child; Female; Fluvoxamine; Human; Male; Serotonin Uptake Inhibitors; Anxiety Disorders -- *drug therapy; Fluvoxamine -- *therapeutic use; Serotonin Uptake Inhibitors -- *therapeutic use
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Anxiety Disorders; Generalized Anxiety Disorder; Phobia, Social; Anxiety, Separation | interventions — Fluvoxamine

INTERVENTIONS:
Drug: Fluvoxamine

SUMMARY:
The purpose of this study is to see if it is effective to treat children with anxiety disorders with fluvoxamine.

Fluvoxamine has been successfully used to treat obsessive-compulsive disorder (OCD) in adults and children. Anxiety disorders other than OCD, such as generalized anxiety disorder, social phobia, or separation anxiety, are very common in youth and are not always responsive to behavioral therapies alone. These disorders may respond to fluvoxamine.

A child will be evaluated for 3 weeks before he/she is assigned randomly (like tossing a coin) to receive either fluvoxamine or an inactive placebo for 8 weeks. After this double-blind phase (neither the child/parents nor the doctor know which treatment is being given), the child will have the option of continuing treatment during a 4-month open-label extension period (both the child/parents and the doctor know which the child is receiving).

A child may be eligible for this study if he/she:

Is 6 to 17 years old and has been diagnosed with an anxiety disorder (i.e., generalized anxiety disorder, social phobia, or separation anxiety).

DETAILED DESCRIPTION:
To evaluate fluvoxamine in the treatment of children and adolescents with anxiety disorders.

Fluvoxamine is a serotonin reuptake inhibitor that is FDA-approved for the treatment of obsessive-compulsive disorder (OCD) in adults and children. Anxiety disorders other than OCD are very common in youth and are not always responsive to psychosocial therapies. Fluvoxamine is an alternative treatment.

After a 3-week period of evaluation, patients meeting study entry criteria are randomized to receive either fluvoxamine or placebo for 8 weeks. After this double-blind phase, patients can enter a 4-month open-label extension.

ELIGIBILITY:
- Patients must have: DSM -IV diagnosis of generalized anxiety disorder, social phobia, or separation anxiety.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 1996-10; Study Completion 1999-11

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Greenhill, MD, Principal Investigator; Mark Riddle, MD, Principal Investigator

REFERENCES:
- [Background] Fluvoxamine for the treatment of anxiety disorders in children and adolescents. The Research Unit on Pediatric Psychopharmacology Anxiety Study Group. N Engl J Med. 2001 Apr 26;344(17):1279-85. doi: 10.1056/NEJM200104263441703. PMID 11323729
- [Background] Coyle JT. Drug treatment of anxiety disorders in children. N Engl J Med. 2001 Apr 26;344(17):1326-7. doi: 10.1056/NEJM200104263441711. No abstract available. PMID 11320394